CLINICAL TRIAL: NCT05902104
Title: CAMP: CGM-Assisted Management of PN
Brief Title: CGM-Assisted Management of PN
Acronym: CAMP
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Agus, Division Chief, Medical Critical Care, Boston Children's Hospital
Other Study IDs: IRB-P00039631
Record Dates: First submitted 2023-05-25; First posted 2023-06-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Intestinal Failure; Hypoglycemia; Hyperglycemia
Keywords: Intestinal Failure; Parenteral Nutrition; Continuous Glucose Monitoring; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Intestinal Failure; Hypoglycemia; Hyperglycemia; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to learn more about changes in glucose levels in hospitalized infants with intestinal failure receiving parenteral nutrition or PN (nutrients delivered intravenously), as they transition from continuous PN (given 24 hours a day) to cycled PN (given less than 24 hours a day).

There is an increased risk of glucose abnormalities with cycled PN, which can be harmful to infant growth and brain health. Continuous glucose monitors (CGM) will be used to measure interstitial glucose levels (in the tissue under the skin), which are similar to blood glucose levels. CGM is a small, minimally-invasive sensor worn on the thigh, which gives a glucose measurement every 5 minutes, and can help us understand changes in blood sugar levels without having to do a blood draw or fingerstick. CGM will be used during PN cycling for up to 30 days or until hospital discharge. If target GIR cycled PN is not reached following 3 sensor periods (up to 10 days per sensor), the parent/guardian will be approached to accept or decline participation in an optional extension phase. In the extension phase, the primary study will be repeated and CGM monitoring will continue until target GIR cycled PN is reached, up to an additional 3 sensor placements. CGM data will be hidden from the clinical team, there will be no change to routine clinical care. CGM may provide false low glucose readings when the tissue around the sensor is compressed (compression lows), such as when laying on the sensor during sleep. We will generate data during the study to help identify and filter the final dataset to remove likely compression lows.

This study may help us understand how cycled PN affects glucose levels in infants with intestinal failure, which may help other children treated with cycled PN in the future.

DETAILED DESCRIPTION:
The objective of this investigation is to quantify dysglycemia associated with cycled parenteral nutrition (PN) and elevated glucose infusion rates (GIR) in infants with intestinal failure and PN-dependence, leveraging high-frequency continuous glucose monitor (CGM) sensor glucose values in a prospective, observational study.

Intestinal failure is a malabsorptive state which necessitates PN in its most severe form. PN is ideally transitioned from continuous (24 hr/day) to cycled PN (<24 hr/day), requiring higher glucose infusion rates (GIR) to provide the same nutrition content over a shorter time-period. Patients on cycled PN, especially infants, are vulnerable to dysglycemia (abnormal glucose levels), specifically hyperglycemia during PN infusions (due to inadequate insulin relative to high GIR) and hypoglycemia when PN is cycled off (due to delayed insulin suppression after PN suspension). There is no established pediatric GIR threshold above which the risk of abnormal glucose levels significantly increases.

While current practice relies on intermittent blood glucose checks, continuous glucose monitors (CGM) measure high-frequency glucose profiles via minimally-invasive sensors, and are capable of precisely detecting clinically-actionable trends that may otherwise go unrecognized. The CGM sensor measures interstitial glucose, an accepted proxy for blood glucose in patients > 2 years old with diabetes or glycemic variability. CGM has been successfully used in infants and can fulfill the need for greater quantitative insight into glucose trends in metabolically and neurologically fragile populations, including infants with intestinal failure.

The investigators hypothesize that during high-GIR, cycled PN: a) trough glucose while PN is suspended is less than normal (statistically defined as 100 mg/dL), and b) average glucose while receiving the target (highest) GIR is greater than normal (statistically defined as 120 mg/dL).

Eligible infants will be identified among hospitalized infants at Boston Children's Hospital and followed by the Home Parenteral Nutrition (HPN) program and the Center for Advanced Intestinal Rehabilitation (CAIR). All enrolled participants will have a Dexcom G6 Pro CGM placed within 1 week prior to the anticipated initiation of PN cycling, and CGM will be worn using blinded mode for up to 30 days until target GIR cycled PN is reached (3 sensors maximum). If target GIR cycled PN is not reached following 3 sensor periods (up to 10 days per sensor), the parent/guardian will be approached to accept or decline participation in an optional extension phase. In the extension phase, the primary study will be repeated and CGM monitoring will continue until target GIR cycled PN is reached, up to an additional 3 sensor placements. No CGM will remain in place at the time of discharge.

The CGM readings will remain blinded to the clinical staff members, no real-time CGM alerts will be provided to the clinical staff. The clinical team will manage PN cycling and clinical blood glucose monitoring as per routine clinical practice. Chart review will occur throughout the study period to abstract necessary information about the participant's medical history and interval clinical events.

An initial CGM data review will be conducted by the research team within 72 hours of each sensor removal. The clinical team will be notified if there were intervals meeting the criteria of sustained sensor readings < 50 mg/dL for greater than or equal to 15 minutes. The clinical team will be provided with the criteria for notification, the date/time stamps associated with those event(s), and information about interpreting CGM readings. We will provide this limited information to the clinical team because sustained CGM sensor readings < 50 mg/dL may signify that the participant is at increased risk for hypoglycemia (blood glucose < 70 mg/dL) on cycled PN. The study protocol does not require any blood glucose measurements or other clinical interventions.

Additionally, CGM may provide false low glucose readings when the tissue around the sensor is compressed (compression lows) such as when laying on the sensor during sleep. During study enrollment, a controlled amount of pressure will be applied to the CGM devices worn by CAMP participants during brief testing periods, which will be used to derive a mathematical model of compression lows in infants. These false low readings will be filtered out of the data for accurate data analysis of true low CGM readings. Specifically, the study team will perform brief tests applying pressure to the CGM device and a force sensor will be used to measure the force being applied to the CGM. Up to 1kg force will be applied to the CGM per attempt. There will be up to 2 attempts to apply force and measure a response per day, 3 days of attempts, 6 attempts total, for no more than 20 minutes per attempt. A successful response is defined as a drop in sensor glucose of at least 15 mg/dL sustained until pressure is released.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intestinal failure with PN dependence
* Hospitalized at Boston Children's Hospital
* Age: 60 days to 18 months
* Corrected gestational age: greater than or equal to 40 weeks
* Weight: greater than or equal to 4kg
* Likely to proceed to PN cycling within the next month, as assessed by the clinical team

Exclusion Criteria:

* Underlying medical conditions or medications that predispose to hypoglycemia or hyperglycemia (e.g. insulin administration, systemic glucocorticoids, hyperinsulinism, adrenal insufficiency, other metabolic diseases)
* Diffuse skin disease such that placement of a CGM sensor would be unsafe or difficult to secure
* Known history of allergy or severe reaction to the adhesive/tape that is used to secure the CGM
* Diffuse body edema that would limit accuracy of CGM sensor
* Poor peripheral perfusion or use of vasoactive agents that would limit accuracy of CGM sensor
* Use of medications that interfere with CGM accuracy (e.g. Hydroxyurea, acetaminophen at more than a maximum dose of 1 g every 6 hours up to 4 g every 24 hours)
* Enrolled in competing clinical trial
* Ward of the state

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inpatients at Boston Children's Hospital (BCH) with intestinal failure dependent on PN followed by the Home Parenteral Nutrition (HPN) and/or Center for Advanced Intestinal Rehabilitation (CAIR) program at BCH.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Trough glucose while PN is suspended | Through study completion, up to 30 days
  For each subject, "trough glucose" will be defined as the lowest sensor glucose value, during the entire study period, that occurs while PN is suspended.
Average glucose while receiving the target GIR | Through study completion, up to 30 days
  For each subject, "average glucose" will be defined as an average of all sensor glucose values recorded while receiving the target GIR. "Target GIR" will be defined as the final GIR prior to discharge home, or highest GIR given during the study period if clinical goal GIR is not reached during the study period.

SECONDARY OUTCOMES:
Measures of dysglycemia | Through study completion, up to 30 days
  Secondary outcomes will further quantify the association between cycled PN and dysglycemia (glucose outside 70 - 150 mg/dL) and will include CGM metrics such as: trough, peak, average, area under curve, time dysglycemic, frequency of dysglycemic events >= 15 minutes, timing of dysglycemic event relative to PN cycling.

CONTACTS AND LOCATIONS:
Overall Officials: Michael SD Agus, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bendorf K, Friesen CA, Roberts CC. Glucose response to discontinuation of parenteral nutrition in patients less than 3 years of age. JPEN J Parenter Enteral Nutr. 1996 Mar-Apr;20(2):120-2. doi: 10.1177/0148607196020002120. PMID 8676529
- [Background] Beltrand J, Colomb V, Marinier E, Daubrosse C, Alison M, Burcelin R, Cani PD, Chevenne D, Marchal CL. Lower insulin secretory response to glucose induced by artificial nutrition in children: prolonged and total parenteral nutrition. Pediatr Res. 2007 Nov;62(5):624-9. doi: 10.1203/PDR.0b013e3181559d5c. PMID 17805200
- [Background] Austhof SI, DeChicco R, Cresci G, Corrigan ML, Lopez R, Steiger E, Kirby DF. Expediting Transition to Home Parenteral Nutrition With Fast-Track Cycling. JPEN J Parenter Enteral Nutr. 2017 Mar;41(3):446-454. doi: 10.1177/0148607115595620. Epub 2016 Sep 29. PMID 26187939
- [Background] Yanagisawa R, Takeuchi K, Komori K, Fujihara I, Hidaka Y, Morita D, Futatsugi A, Ono T, Hidaka E, Sakashita K, Shiohara M. Hypoglycemia During the Temporary Interruption of Parenteral Nutrition Infusion in Pediatric Hematopoietic Stem Cell Transplantation. JPEN J Parenter Enteral Nutr. 2017 Nov;41(8):1414-1418. doi: 10.1177/0148607116665797. Epub 2016 Aug 23. PMID 27554675